CLINICAL TRIAL: NCT00247442
Title: An Evaluation of a Decision Aid for Women Aged Over 70 Considering Whether to Stop or Continue Having Mammography Screening.
Brief Title: Australian Screening Mammography Decision Aid Trial (ASMDAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CD-9999999
Record Dates: First submitted 2005-10-30; First posted 2005-11-01 (Estimated); Last update posted 2006-09-28 (Estimated); Status verified 2005-06

CONDITIONS: Breast Neoplasms
Keywords: Mammography screening; Breast cancer screening; Screening outcomes; Decision aid; Decision support tool; Informed choice
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

INTERVENTIONS:
Behavioral: Decision aid

SUMMARY:
The purpose of the study is to develop and evaluate a decision aid to assist women aged 70 years and over to make an informed choice about whether to continue screening mammography.

DETAILED DESCRIPTION:
The primary aims of the study are to assess the impact of the decision aid on (1) the proportion of women who make an informed choice about whether to continue screening mammography, and (2) the participation rates of screening among women aged 70 years and older.

There are two secondary aims of the study. First, to measure the effect of the decision support tool on women's decisional conflict, anxiety, and knowledge about the issues involved in screening mammography. Second, to compare relationships between a woman's objective and perceived risk of breast cancer with her decision to continue or stop screening mammography.

Screening mammography is recommended for women aged 50-69 years but there is no recommendation for women aged 70 years and older. Therefore the decision to continue or stop having screening mammograms are largely dependent on the importance women place on the perceived benefits and harms of screening.

The decision aid is a paper workbook and worksheet containing information on the outcomes of screening mammography for women aged 70 years and older (based on a published model- Barratt et al. 2005), steps to decision making and values clarification exercise. Currently it is not known if a decision aid with information about the benefits and risks of screening mammography can help women aged 70 years and older to make an informed choice. In addition to delivering benefits to individual women in assisting them to to make an informed choice the decision aid may lead to benefits for service providers such as improved efficiency and cost-effectiveness of screening women in this age group. Thus the impact of a decision aid in the efficiency and cost-effectiveness of screening mammography is an important but untested hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Women who are due their FIRST screening mammogram over the age of 70, and who have previously participated in screening mammography at BreastScreen NSW.

Exclusion Criteria:

* Inability to complete a telephone interview in English.
* Personal history of breast cancer (invasive and pre-invasive).

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 670
Dates: Start 2006-01; Study Completion 2006-04

PRIMARY OUTCOMES:
Informed choice
Participation

SECONDARY OUTCOMES:
Decisional conflict
Knowledge
Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Heather Davey, B.Psych, MPH, Principal Investigator — University of Sydney; Nehmat Houssami, MBBS, PhD, Principal Investigator — University of Sydney; Erin Mathieu, B.Ed, MPH, Principal Investigator — University of Sydney; Andrew Page, BA (Hons), Principal Investigator — BreastScreen NSW; Richard Taylor, MBBS, PhD, Principal Investigator — BreastScreen NSW; Sian Smith, BSc (Hons), Principal Investigator — University of Sydney; Phyllis Butow, MPH, PhD, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Riganti P, Ruiz Yanzi MV, Escobar Liquitay CM, Sgarbossa NJ, Alarcon-Ruiz CA, Kopitowski KS, Franco JV. Shared decision-making for supporting women's decisions about breast cancer screening. Cochrane Database Syst Rev. 2024 May 10;5(5):CD013822. doi: 10.1002/14651858.CD013822.pub2. PMID 38726892